CLINICAL TRIAL: NCT02270346
Title: Effects of Inspiratory Muscle Training in Allogeneic Hematopoietic Stem Cell Transplantation Recipients
Brief Title: Inspiratory Muscle Training in Allogeneic Hematopoietic Stem Cell Transplantation Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Assoc. Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GaziUniversity
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Allogeneic HSCT, Inspiratory Muscle Training, Exercise Capacity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): Intervention: Treatment group received inspiratory muscle training (IMT) using POWERbreathe Classic threshold loading device.
  Interventions: Device: Inspiratory muscle training
- Control group (Sham Comparator): Sham: Control group received sham inspiratory muscle training (IMT) using POWERbreathe Classic threshold loading device .
  Interventions: Device: Sham inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — Treatment group received inspiratory muscle training using threshold loading device (POWERbreathe Classic, IMT Technologies Ltd. Birmingham, England) at 40% of maximal inspiratory pressure (MIP).
  The MIP was measured at supervised session each week, and 40% of measured MIP value was the new training workload.
  The treatment group trained for 30 min-per/day, 7 days/week, for 6 weeks. Six sessions at home and 1 session were performed at department.
  Arms: Treatment group
Device: Sham inspiratory muscle training — Control group received sham inspiratory muscle training using threshold loading device (POWERbreathe Classic IMT Technologies Ltd. Birmingham, England) at fixed workload, 5% of MIP.
  The control group trained for 30 min-per/day, 7 days/week, for 6 weeks. Six sessions at home and 1 session were performed at department.
  Arms: Control group

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) causes various toxic effects in many body tissues, organs and systems such as immune, cardiovascular, pulmonary, gastrointestinal, neuroendocrine and musculoskeletal systems, liver, kidneys and skin.Available limited numbers of studies showed that inspiratory muscle weakness in allo-HSCT candidates and recipients. Although meta-analysis, systematic reviews and studies demonstrated beneficial effects of inspiratory muscle training on several outcomes in different disease groups; chronic obstructive pulmonary disease, bronchiectasis and heart failure, no published paper reported the effects of IMT in allo-HSC recipients.

DETAILED DESCRIPTION:
Thirty-eight allo-HSCT recipients (˃100 days past post-transplant status) were included. Before and after 6-week IMT, maximal and submaximal exercise capacity, respiratory and peripheral muscle strength, pulmonary functions, dyspnea and fatigue perception, depression and quality of life were evaluated. Primary outcome measurement was respiratory muscle strength, secondary outcomes were exercise capacity, dyspnea, peripheral muscle strength, quality of life, fatigue and depression.

ELIGIBILITY:
Inclusion Criteria:

* Allo-HSC recipients (˃100 days past post-transplant status),
* 18-65 years of age,
* Under standard medications

Exclusion Criteria:

* Having cognitive disorder, orthopedic problem or neurological disease that were affecting functional capacity,
* Additional heart and lung diseases such as asthma, chronic obstructive pulmonary disease, acute infections or pneumonia,
* Problems prevented performing assessment and training such as visual problems and mucositis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Inspiratory and expiratory muscle strength (MIP, MEP) | 6 weeks
  Mouth pressure device

SECONDARY OUTCOMES:
Fatigue | 6 weeks
  Fatigue Impact Scale (FIS)
Pulmonary function | 6 weeks
  Spirometry
Peripheral muscle strength | 6 weeks
  Hand held dynamometer
Dyspnea | 6 weeks
  Modified Borg and Modified Medical Research Council (MMRC) dyspnea scales,
Depression | 6 weeks
  Montgomery Asberg Depression Rating Scale (MADRS)
Quality of life | 6 weeks
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C-30 version 3.0 (Turkish versions of all scales)
Submaximal exercise capacity | 6 weeks
  Six-minute walk test (6MWT)
Maximal exercise capacity | 6 weeks
  Modified incremental shuttle walk test (ISWT)

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, MSc., Study Chair — Gazi University; Meral Boşnak Güçlü, PhD., Study Director — Gazi University; Zeynep Arıbaş, MSc., Principal Investigator — Gazi University; Zeynep Şahika Akı, MD, PhD., Principal Investigator — Gazi University; Gülsan Türköz Sucak, MD, PhD., Principal Investigator — Gazi University

REFERENCES:
- [Result] Dimeo FC, Tilmann MH, Bertz H, Kanz L, Mertelsmann R, Keul J. Aerobic exercise in the rehabilitation of cancer patients after high dose chemotherapy and autologous peripheral stem cell transplantation. Cancer. 1997 May 1;79(9):1717-22. PMID 9128987
- [Result] Ferrell B, Grant M, Schmidt GM, Rhiner M, Whitehead C, Fonbuena P, Forman SJ. The meaning of quality of life for bone marrow transplant survivors. Part 1. The impact of bone marrow transplant on quality of life. Cancer Nurs. 1992 Jun;15(3):153-60. PMID 1611601
- [Result] White AC, Terrin N, Miller KB, Ryan HF. Impaired respiratory and skeletal muscle strength in patients prior to hematopoietic stem-cell transplantation. Chest. 2005 Jul;128(1):145-52. doi: 10.1378/chest.128.1.145. PMID 16002928
- [Result] Kovalszki A, Schumaker GL, Klein A, Terrin N, White AC. Reduced respiratory and skeletal muscle strength in survivors of sibling or unrelated donor hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Jun;41(11):965-9. doi: 10.1038/bmt.2008.15. Epub 2008 Feb 11. PMID 18264142
- [Derived] Bargi G, Guclu MB, Aribas Z, Aki SZ, Sucak GT. Inspiratory muscle training in allogeneic hematopoietic stem cell transplantation recipients: a randomized controlled trial. Support Care Cancer. 2016 Feb;24(2):647-659. doi: 10.1007/s00520-015-2825-3. Epub 2015 Jul 2. PMID 26135532